CLINICAL TRIAL: NCT06841731
Title: A Multi-center, Randomized, Double-blind, Active Controlled, Parallel Groups, Phase II Study to Evaluate the Efficacy and Safety of HRS-8427 in the Treatment of Adults With Hospital-acquired Bacterial Pneumonia (HABP) or Ventilator-associated Bacterial Pneumonia (VABP)
Brief Title: A Trial of HRS-8427 in the Treatment of Adults With Bacterial Pneumonia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-8427-201
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Hospital-acquired Bacterial Pneumonia (HABP); Ventilator-associated Bacterial Pneumonia (VABP)
MeSH Terms: interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-8427 (Experimental)
  Interventions: Drug: HRS-8427
- Meropenem (Active Comparator)
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: HRS-8427 — HRS-8427 for injection.
  Arms: HRS-8427
Drug: Meropenem — Meropenem for injection.
  Arms: Meropenem

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of HRS -8427 in patients with HABP/VABP.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide a written informed consent before the study, fully understand the study and be able to complete the study according to the protocol.
2. Male and female, ≥18 years.
3. Judged by the investigator, clinical diagnosis with HABP/VABP, expectation that the patients will require hospitalization and initial treatment with intravenous antibiotics.
4. All subjects must have a chest radiograph during screening or within 48h before randomization, showing the presence of new or progressive infiltrate(s) suggestive of bacterial pneumonia.
5. Women of childbearing potential must have a negative serum pregnancy test before the first dose and must be non-lactating. Fertile female subjects or male subjects whose partner is a fertile female agree to use highly effective form of contraception, with no plan of birth and sperm/ovum donation from the time of signing the informed consent form (ICF) till 14 days after the end of treatment.

Exclusion Criteria:

1. Subjects who have known or suspected community-acquired bacterial pneumonia (CABP), atypical pneumonia, or chemical pneumonia.
2. Subjects who have known or suspected pneumonia caused by mycoplasma, chlamydia, legionella, viruses, fungi or parasites.
3. HABP or VABP caused by obstruction.
4. Subjects who have received potentially effective antibiotic therapy for a continuous duration of more than 24 hours during the previous 72 hours prior to randomization.
5. Impairment of renal function with estimated glomerular filtration rate < 15 mL/min, or receiving peritoneal dialysis/hemodialysis.
6. Subjects with significant laboratory abnormalities.
7. Other pulmonary diseases that may confound the assessment of efficacy or safety.
8. Known history of immune deficiency disease or receive immunocompromising treatment.
9. Severe cardiovascular and cerebrovascular diseases with clinical significance and unstable or uncontrolled condition.
10. Known or suspected central nervous system infections.
11. Patients received cancer treatment within 4 weeks before randomization or planned treatment during the study period.
12. Drug abuse within 1 year prior to randomization.
13. Judged by the Investigator, other reasons unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The all-cause mortality rate at Day 14. | From the first dose of the study drug to Day 14.

SECONDARY OUTCOMES:
The all-cause mortality rate at Day 28. | From the first dose of the study drug to Day 28.
The total ventilation time. | Day 14 to Day 21.
The total ventilation time. | Day 21 to Day 28.
The percentage of participants with microbiologic eradication at the early assessment (EA) period. | Day 4 after the start of the treatment.
The percentage of participants with microbiologic eradication at the end of treatment (EOT) period. | Day 7 to 14.
The percentage of participants with microbiologic eradication at the test of cure (TOC) period. | Day 14 to 21.
The percentage of participants with microbiologic eradication at the follow-up (FU) period. | Day 21 to 28.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided